CLINICAL TRIAL: NCT03957239
Title: The Effect of a Cranberry Beverage on Intestinal Permeability and Gastrointestinal Function in Generally Healthy Adults With a BMI ≥ 30: a Randomized, Double-blind, Controlled, Crossover Study
Brief Title: The Effect of a Cranberry Beverage on Intestinal Permeability and Gastrointestinal Function in Generally Healthy Adults
Acronym: MAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201901253; OCR21702 (Other: UF OnCore)
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Intestinal Permeability; Gastrointestinal Function

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled crossover in which participants receive one of the study beverages (cranberry or cranberry-flavored) for a 2-week intervention period each will be used.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, investigators, and anyone else involved with the study will remain blinded for its entirety.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry Beverage (Experimental): Four prepackaged juice boxes (4.23 oz each) containing a whole milled cranberry beverage for 2 weeks
  Interventions: Other: Cranberry Beverage
- Placebo Group (Placebo Comparator): Four prepackaged juice boxes (4.23 oz each) containing a cranberry-flavored beverage for 2 weeks
  Interventions: Other: Control Beverage

INTERVENTIONS:
Other: Cranberry Beverage — The cranberry beverage will provide 50 kcals and 4.0 grams of fiber per day from whole milled cranberries, water, cranberry natural flavor and sucralose.
  Arms: Cranberry Beverage
Other: Control Beverage — The control beverage will provide 50 kcals per day and is a color, taste matched sugar sweetened beverage formulated with water, sucrose, citric acid, cranberry natural flavor, malic acid, xanthum gum, sucralose and artificial color (red 40, blue 1).
  Arms: Placebo Group

SUMMARY:
In this double blind, crossover study participants will consume a cranberry beverage and a cranberry-flavored beverage for 2 weeks each. Gut permeability will be assessed weekly using aspirin and food-grade sugar molecules. Participants will be asked to provide urine, blood, saliva and stool samples to assess gut permeability and microbial communities. No change in permeability to the small sugar probes is anticipated with the cranberry beverage

DETAILED DESCRIPTION:
Obesity, stress, liver disease, alcoholism, diabetes, and autoimmune diseases in humans or animal models are associated with altered intestinal permeability; consequently, maintenance of the gastrointestinal barrier is an emerging area of interest. The purpose of this randomized, double-blind, controlled crossover study is to compare the difference between the change from baseline in gastroduodenal permeability after drinking a cranberry or control beverage for two weeks. Gastroduodenal permeability will be assessed following aspirin challenge by measuring urinary sucrose in the 0 to 5-hour urine collection after differential sugar probes are consumed. Urine will be collected for an additional 19 hours (24 hours total) to assess whole gut permeability. A 4-week washout period will separate the interventions. Stool and fasting blood and saliva samples will be obtained before and during the intervention periods to assess fecal microbial communities and markers of intestinal barrier, immune function and oxidative stress. It is anticipated that cranberry juice will selectively increase intestinal Akkermansia bacteria, reduce markers of inflammation and oxidative stress, increase mucosal immunity, and protect the gastroduodenal barrier from an aspirin challenge.

ELIGIBILITY:
Inclusion Criteria

* Have a BMI ≥ 30 kg/m2 and a waist circumference ≥ 35 inches for women and ≥ 40 inches for men.
* Have had a stable weight for 3 months (<5 kg or ~11 lbs body weight change)
* Willing to discontinue the use of non-steroidal anti-inflammatory drugs (NSAIDs), such as ibuprofen, aspirin, naproxen, or indomethacin, for the full length of the study.
* Willing to discontinue consumption of wine and berries throughout the 12-week study.
* Willing and able to avoid consumption of any cranberry juice, whole cranberries, and dried cranberries during the two weeks leading up to the study and during the study, not including the study beverage.
* Willing to avoid beer and cocktails on the day before and the day of the sugar probe tests.
* Willing to avoid the use of antidiarrheal or laxative medication on a regular or an "as-needed basis" during the full length of the study.
* Willing to provide urine, saliva, blood, and stool samples during the study collection periods.
* Have used aspirin in the past and did not experience adverse effects.
* Willing to consume three tablets (325 mg each or 975 mg total) twice within a 9 to 12-hour period. This challenge will be repeated four times during the 12-week study.
* Willing and able to complete daily and weekly questionnaires online regarding dietary intake and general health and well-being, including gastrointestinal habits.
* Willing to discontinue consumption of fermented foods or probiotics.
* Willing to discontinue consumption of fiber supplements.
* Willing to discontinue taking prebiotic, herbal, or high-dose vitamin or mineral supplements that may impact immune function or inflammation during the pre-baseline period and throughout the study protocol.
* Willing and able to consume 4.23 oz of a cranberry beverage four times daily (~16 oz total/d) for the 2-week study interventions.
* Willing to avoid high intensity exercises two days prior to and the day of the permeability tests. These tests will be done on four occasions.
* Willing and able to complete the informed consent form in English.
* Willing to provide a social security number to receive study payment.

Exclusion Criteria

* Currently being treated for a physician-diagnosed gastrointestinal disease or condition (such as ulcerative colitis, Crohn's disease, gastroparesis, cancer, peptic ulcer disease, Celiac disease, short bowel disease, ileostomy, or colostomy) other than GERD or diverticular disease
* Currently being treated for or type 1 diabetes or type 2 diabetes by medication
* Daily use of NSAIDs in the last 3 months or incidental use in the last 2 weeks prior to screening.
* Allergy to aspirin or cranberries.
* Participate in moderate or high exercise activities during a typical week.
* Currently smoking (including vaping) tobacco products
* Women who are lactating, pregnant, or are attempting to get pregnant.
* Use of another investigational product within 3 months of the screening visit.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Change in Gastroduodenal permeability | Baseline and Week 2 of each intervention
  Compare the statistical difference between the change from baseline (i.e., final - baseline) in gastroduodenal permeability after consuming the cranberry beverage for 2 weeks versus the change after consuming the control beverage for 2 weeks. Gastroduodenal permeability will be assessed following aspirin challenge by measuring urinary sucrose in the 0 to 5-hour urine collection.

SECONDARY OUTCOMES:
Change in Small intestinal permeability | Baseline and Week 2 of each intervention
  Compare the difference between the changes in lactulose/rhamnose concentrations in a 5-hour urine collection (end of intervention minus baseline) from the cranberry beverage versus control beverage
Change in Colonic permeability | Baseline and Week 2 of each intervention
  Compare the difference between the changes in sucralose/ erythritol ratio in the 5 to 24-hour urine collection (end of intervention minus baseline) from the cranberry beverage vs control beverage
Change in Whole gut permeability | Baseline and Week 2 of each intervention
  Compare the difference between the changes in sucralose/ erythritol ratio in the 0 to 24-hour urine collection (end of intervention minus baseline) from the cranberry beverage vs control beverage
Change in Stool consistency | Baseline and Week 2 of each intervention
  Compare the average stool consistency (Bristol Stool Form Scale) between the cranberry beverage versus control beverage. The Bristol Stool Form Scale (BSS) measures stool types from 1-7 with 1 = hard and 7 = liquid. A score from 3-5 is indicative of a normal BSS.
Change in Stool frequency | Baseline and Week 2 of each intervention
  Compare the number of number of stools between the cranberry beverage versus control beverage
Change in Bacterial species of interest | Baseline and Week 2 of each intervention
  Compare the genome equivalents between the cranberry beverage versus control beverage. Genome equivalents will be measured by quantitative polymerase chain reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No